CLINICAL TRIAL: NCT01173211
Title: A Randomized, Double-Blind Trial on the Safety and Immunogenicity of Seasonal 2010-2011 Inactivated Trivalent Influenza Vaccine in Pregnant Women
Brief Title: 2010-2011 Trivalent Influenza Vaccine (TIV) in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0005; HHSN272200800002C
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2013-03

CONDITIONS: Influenza
Keywords: pregnant, women, influenza, vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Arm 1: Fluarix® (Experimental): 60 pregnant women and 20 non-pregnant women to receive a single intramuscular 0.5 mL dose of Fluarix®.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Arm 3: Fluzone® (Experimental): 60 pregnant women and 20 non-pregnant women to receive a single intramuscular 0.5 mL dose of Fluzone®.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Arm 2: Agriflu® (Experimental): 60 pregnant women and 20 non-pregnant women to receive a single intramuscular 0.5 mL dose of Agriflu®.
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Three licensed 2010-2011 seasonal inactivated trivalent influenza vaccines. Single intramuscular 0.5 mL dose. Each vaccine is formulated to contain 45 micrograms (mcg) hemagglutinin (HA) per 0.5 mL dose. Thimerosal is a preservative used in some vaccines. Fluzone, Agriflu and Fluarix do not contain thimerosal. For Fluarix, the tip cap and rubber plunger of the needleless prefilled syringes contain dry natural latex rubber.
  Arms: Arm 2: Agriflu®
Biological: Trivalent inactivated influenza vaccine — Three licensed 2010-2011 seasonal inactivated trivalent influenza vaccines. Single intramuscular 0.5 mL dose. Each vaccine is formulated to contain 45 micrograms (mcg) hemagglutinin (HA) per 0.5 mL dose. Thimerosal is a preservative used in some vaccines. Fluzone, Agriflu and Fluarix do not contain thimerosal. For Fluarix, the tip cap and rubber plunger of the needleless prefilled syringes contain dry natural latex rubber..
  Arms: Arm 3: Fluzone®
Biological: Trivalent inactivated influenza vaccine — Three licensed 2010-2011 seasonal inactivated trivalent influenza vaccines. Single intramuscular 0.5 mL dose. Each vaccine is formulated to contain 45 micrograms (mcg) hemagglutinin (HA) per 0.5 mL dose. Thimerosal is a preservative used in some vaccines. Fluzone®, Agriflu® and Fluarix® do not contain thimerosal. For Fluarix, the tip cap and rubber plunger of the needleless prefilled syringes contain dry natural latex rubber.
  Arms: Arm 1: Fluarix®

SUMMARY:
The purpose of this study is to see how much antibody (proteins produced by the immune system that help fight infections) the body makes after getting a flu vaccine. Researchers will also look at how the body reacts to the flu vaccine and how it affects the babies of pregnant women. The study will enroll approximately 240 women ages 18-39 years, including 180 pregnant women in their second or third trimester of pregnancy (at least 14 weeks pregnant) and 60 non-pregnant women. Participants will be randomly (by chance) assigned to 1 of 3 vaccine groups. Each participant will receive one shot of a 2010-2011 flu season licensed vaccine. The vaccine will be given as an intramuscular injection (shot in the muscle) in the upper arm. Study procedures include pregnancy testing, blood draws, and memory aids. Patient participation may be up to 8 months. The information from this study will help guide researchers in developing flu vaccines for pregnant women.

DETAILED DESCRIPTION:
Influenza is a significant cause of morbidity and mortality in the United States. Pregnant women and infants are at an increased risk for the complications of influenza. Pregnant women are considered a high risk population. In the United States, routine vaccination with inactivated trivalent influenza vaccine (TIV) for women who are pregnant or deliver during the influenza season is recommended. However, few studies exist on the safety and immunogenicity of administration of seasonal inactivated TIV. Although influenza vaccination has been recommended during pregnancy, the rates of immunization remain low, at about 13 percent, which partly reflects concern of safety among pregnant women and providers. It is important to gather prospective data on the safety and immunogenicity of inactivated TIV vaccine in pregnant women. This is a multi-site randomized, double-blinded clinical trial in 180 healthy 18-39 year old, pregnant women in their second or third trimester of pregnancy (from 14 weeks of gestation to 33 weeks/6 days gestation, inclusive) and 60 healthy 18-39 year old non-pregnant controls. Study subjects will be randomized 1:1:1 to receive one of the following three 2010-2011 seasonal inactivated trivalent influenza vaccines: Fluarix®, Agriflu®, or Fluzone® (60 pregnant women and 20 non-pregnant women per group). The study will begin enrollment when at least 2 of the 4 study products are available. Once enrolled, a blood sample will be collected and each subject will receive a single 0.5 mL dose of the assigned vaccine. Subjects will be observed for at least 15 minutes after immunization, and the subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 8 days after immunization. Subjects will have a phone call on Day 2 and 8 for review of memory aid, concomitant medication assessment, and assessment of AEs. At approximately Day 28 post-vaccination, subjects will return to the clinic for blood sample collection, AE and concomitant medication assessment, and a targeted physical examination (if indicated). Pregnant subjects will also have scheduled phone calls from Day 28 until the time of delivery or Day 180, whichever is later, to assess for any new-onset chronic medical conditions, and pregnancy-related problems such as miscarriage or serious adverse events (SAEs) since the last visit. At approximately Day 180 post-vaccination, subjects will return to the clinic for blood sample collection and assessment of the receipt of any vaccines since the last visit. Subjects will be asked about any new-onset chronic medical conditions, SAEs since the last visit and pregnancy-related problems such as miscarriage (for the pregnant women cohort). The duration of the study will be approximately 6 months for the non-pregnant subjects and about 6-8 months for the pregnant subjects, depending on delivery date for the pregnant women. Pregnant subjects will have collection of maternal and cord blood at the time of delivery. Pregnant subjects will also have a phone call 1 month after delivery to assess for any new-onset chronic medical conditions or SAEs since the last visit. The primary objectives are to evaluate the safety of a single 0.5 mL intramuscular injection of the 2010-2011 inactivated TIV in pregnant women and to evaluate the immunogenicity of the 2010-2011 inactivated TIV in pregnant women by hemagglutination inhibition assay (HAI). The secondary objectives are to evaluate the persistence of antibodies to the 2010-2011 inactivated TIV in pregnant women at Day 180 and to assess the transfer of maternally derived antibody against viruses in the 2010-2011 inactivated TIV to infants bor

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

* Pregnant female between the ages of 18 and 39 years, inclusive.
* Is a singleton pregnancy and is from 14 weeks/0 days through 33 weeks/6 days of gestation.
* Had at least one prenatal visit during which pregnancy was confirmed.
* Is in good health, as determined by vital signs [heart rate <100 beats per minute (bpm); blood pressure: systolic <140 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature <100 degrees Fahrenheit], medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history. A stable medical condition is defined as health outcomes of a specific disease are considered to be within acceptable limits in the last 3 months.
* Intends to be available through 6 months following receipt of 2010-2011 seasonal influenza vaccine or until all delivery record information has been obtained, whichever is longer.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.
* Agrees to sign medical release for herself and her infant to allow study staff to gather pertinent medical information and pregnancy outcome data, if needed per clinical site policy.

Non-pregnant women:

* Female between the ages of 18-39 years, inclusive.
* For the 30 days prior to enrollment through 30 days following receipt of 2010-2011 inactivated trivalent influenza vaccine (TIV) in the study must fulfill one of the following: (i) she is not able to bear children because she has been surgically sterilized (hysterectomy) or is at least 1 year status post tubal ligation or 1 year post-menopausal or (ii) she agrees to practice effective methods of contraception including, but not limited to, abstinence, barrier methods (such as a condom or diaphragm) used with a spermicide, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices), or monogamy with vasectomized partner.
* For a female subject of childbearing potential, must have a negative pregnancy test (urine or serum) within 24 hours prior to vaccination.
* Is in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history (if indicated). A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
* Intends to be available through 6 months following receipt of 2010-2011 inactivated TIV.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.

Infants born to pregnant women:

* Infant aged 6 weeks (plus/minus 14 days), born to mothers enrolled in this study.
* Had a cord blood sample collected at time of labor and delivery.
* Parent(s)/legal guardian(s) must be willing and able to comply with planned study procedures and be available for study visit.
* Subject and/or parent(s)/legal guardian(s) must provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

Pregnant women:

* Has received the 2010-2011 trivalent influenza vaccine (inactivated or live).
* Has a known allergy or hypersensitivity to eggs, egg proteins, latex or other components in the vaccines (including, but not limited to: formaldehyde, polyethylene glycol p-isooctylphenyl ether, sucrose, gelatin, polysorbate 80, kanamycin, polymyxin and neomycin).
* Has a history of severe reactions following previous immunization with influenza virus vaccines.
* Has received any other live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 28 days following vaccination. Measles, mumps, and rubella vaccine and tetanus, diphtheria, and acellular pertussis vaccine and human papillomavirus vaccine are permitted post-partum.
* Is enrolled or plans to enroll in another interventional clinical trial with an investigational product during the current pregnancy and while participating in this study (observational studies are allowed).
* Has an acute illness and/or an oral temperature >/= 100.0 degrees F, within 72 hours of vaccination (This may result in a temporary delay of vaccination).
* Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants (a daily aspirin may be acceptable).
* Long term use of glucocorticoids, including oral or parenteral, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed) or has received betamethasone or dexamethasone to accelerate fetal lung maturity.
* Has a history of receiving immunoglobulin or other blood product (with exception of Rhogam) within the 3 months prior to enrollment in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* The subject is receiving any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving an antidepressant drug (not listed above) and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of alcohol or drug abuse in the last 5 years.
* Has a seizure disorder or is on an anti-seizure medication.
* Has a history of Guillain-Barré Syndrome.
* Has an acute or chronic medical condition that, in the opinion of the investigator would render vaccination unsafe, or would interfere with the evaluation of responses (this includes, but is not limited to, known cardiac disease, chronic hypertension, chronic liver disease, significant renal disease, unstable or progressive neurological disorder, transplant recipients or diabetes, juvenile diabetes [Type I] or advanced diabetes with renal disease or eye disease. Gestational diabetes controlled by diet or insulin is acceptable).
* Has any of the following active medical conditions at the time of enrollment:

Hyperemesis gravidarium, premature labor (regular uterine contractions with cervical change), fetus with known major congenital anomaly or genetic abnormality, fetal growth restriction, preeclampsia, or known uterine anomaly (e.g. bicornuate uterus, submucosal fibroids > 5cm).

* Has a history of preeclampsia or preterm birth <35 weeks gestation during a previous pregnancy
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Non-pregnant women:

* Has received the 2010-2011 trivalent influenza vaccine (inactivated or live).
* Has a known allergy or hypersensitivity to eggs, egg proteins, latex or other components in the vaccines (these may include, but not limited to: formaldehyde, polyethylene glycol p-isooctylphenyl ether, sucrose, gelatin, polysorbate 80, kanamycin, polymyxin and neomycin).
* Has a history of severe reactions following previous immunization with influenza virus vaccines.
* Has received any other live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 28 days following vaccination.
* Is enrolled or plans to enroll in another interventional clinical trial with an investigational product at the time of enrollment or during participation in this trial (observational studies are allowed).
* Has an acute illness and/or an oral temperature greater than or equal to 100.0 degrees F, within 72 hours of vaccination (This may result in a temporary delay of vaccination).
* Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants (daily aspirin may be acceptable.
* Long term use of glucocorticoids, including oral or parenteral, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* The subject is receiving any of the following psychiatric drugs: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. Subjects who are receiving an antidepressant drug (not listed below) and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Known active infection with HIV, hepatitis B, or hepatitis C.
* History of alcohol or drug abuse in the last 5 years.
* Has a seizure disorder or is on an anti-seizure medication.
* Has a history of Guillain-Barré Syndrome.
* Has an acute or chronic medical condition that, in the opinion of the investigator would render vaccination unsafe, or would interfere with the evaluation of responses (this includes, but is not limited to, known cardiac disease, chronic liver disease, significant renal disease, unstable or progressive neurological disorder, transplant recipients or uncontrolled diabetes, juvenile diabetes [Type I] or advanced diabetes with renal disease or eye disease. Diabetes controlled by diet or oral agents is acceptable).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Infants born to pregnant women:

- Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke University Medical Center - Duke Perinatal Clinic, Durham, North Carolina
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy pregnant women recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 28Sep2010 and 27Apr2011
Groups:
- Agriflu (Novartis) in Pregnant Participants: Participants in their second or third trimester of pregnancy received a single intramuscular injection of Agriflu (manufacturer Novartis), 45 mcg total antigen per dose
- Fluarix (GSK) in Pregnant Participants: Participants in their second or third trimester of pregnancy received a single intramuscular injection of Fluarix (manufacturer GSK), 45 mcg total antigen per dose
- Fluzone (Sanofi Pasteur) in Pregnant Participants: Participants in their second or third trimester of pregnancy received a single intramuscular injection of Fluzone (manufacturer sanofi pasteur), 45 mcg total antigen per dose
- Agriflu (Novartis) in Non-pregnant Participants: Non-pregnant participants received a single intramuscular injection of Agriflu (manufacturer Novartis), 45 mcg total antigen per dose
- Fluarix (GSK) in Non-pregnant Participants: Non-pregnant participants received a single intramuscular injection of Fluarix (manufacturer GSK), 45 mcg total antigen per dose
- Fluzone (Sanofi Pasteur) in Non-pregnant Participants: Non-pregnant participants received a single intramuscular injection of Fluzone (manufacturer sanofi pasteur), 45 mcg total antigen per dose
Period: Overall Study
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Started | 48 | 45 | 46 | 15 | 16 | 13
Completed | 46 | 44 | 44 | 15 | 16 | 13
Not Completed | 2 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants | Total
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 45 | 46 | 15 | 16 | 13 | 183
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (4.4) | 29.8 (4.1) | 30.7 (4.8) | 27.5 (6.5) | 29.3 (6.7) | 29.7 (5.2) | 30.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 46 | 15 | 16 | 13 | 183
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 46 | 15 | 16 | 13 | 183

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Vaccine-associated Unsolicited Non-serious Adverse Events
Description: Unsolicited non-serious adverse events were collected from participants at follow up contacts, either by phone or in clinic, through 28 days after vaccination. Association to vaccination was determined by a clinician licensed to make a medical diagnosis and listed on the site's Federal Drug Administration's Form 1572.
Time Frame: Day 0 through Day 28 post vaccination
Population: All participants receiving vaccination are included in the safety cohort
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants | 2 | 3 | 2 | 0 | 1 | 1

2. Primary Outcome: Number of Participants Reporting Maternal Complications of Pregnancy, Labor and Delivery
Description: Participants were contacted after delivery, and medical records reviewed, to collect complications experienced during pregnancy, labor and delivery. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: During the pregnancy and at the time of delivery
Population: Pregnant participants receiving vaccination are included in this outcome measure.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46
participants
  Stillborn | 0 | 0 | 0
  Miscarriage | 0 | 0 | 0
  Gestational Diabetes | 2 | 2 | 2
  Polyhydramnios | 1 | 0 | 2
  Oligohydramnios | 3 | 3 | 2
  Pregnancy induced hypertension | 3 | 4 | 1
  Pre-eclampsia | 0 | 1 | 0
  Eclampsia | 0 | 0 | 0
  Fetal distress | 5 | 2 | 2
  Abruptio placenta | 0 | 0 | 1
  Chorioamnionitis | 0 | 1 | 1
  Fever greater than 100.4 degrees Fahrenheit | 3 | 2 | 2
  Anaphylaxis | 0 | 0 | 0
  Antibiotics prior to delivery | 23 | 19 | 20
  Fetal abnormalities detected during pregnancy | 5 | 0 | 1
  Other complications during pregnancy or delivery | 26 | 28 | 30
  Assisted vaginal delivery | 3 | 4 | 2
  Non-elective Cesarean section | 6 | 3 | 7
  Abnormal amniotic fluid | 6 | 11 | 13
  Postpartum fever greater than 100.4 degrees Fahren | 2 | 1 | 1
  Postpartum endometritis | 0 | 0 | 0
  Postpartum bleeding | 2 | 3 | 3
  Postpartum bacteremia | 0 | 0 | 0
  Other postpartum complications | 3 | 1 | 7

3. Primary Outcome: Number of Participants Reporting Neonatal Complications
Description: Participants were contacted after delivery, and medical records reviewed, to collect neonatal complications. The data collection process followed a prospectively-defined list of complications reported for this outcome measure, some of which may have also been reported as serious adverse events if otherwise meeting those requirements.
Time Frame: At time of delivery
Population: Pregnant participants receiving vaccination are included in this outcome measure.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46
participants
  Pre-term (less than 37 weeks) | 2 | 4 | 3
  Large for gestational age | 6 | 3 | 8
  Small for gestational age | 2 | 1 | 1
  Abnormal infant exam | 5 | 5 | 11
  Congenital abnormalities | 5 | 0 | 3
  Hematological complications | 3 | 3 | 4
  Infection | 0 | 0 | 2
  Sepsis | 0 | 0 | 0
  Meningitis | 0 | 0 | 0
  Metabolic complications | 2 | 0 | 0
  Respiratory complications | 8 | 7 | 7
  Respiratory support used | 6 | 5 | 6
  Fever greater than 100.4 degrees Fahrenheit | 0 | 1 | 2
  Admission to special nursery/infant intensive care | 4 | 4 | 4
  Other clinical problems | 6 | 5 | 4

4. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death of the mother, fetus or infant; was life threatening to mother, fetus or infant; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; was a congenital anomaly/birth defect in fetus or infant; or may have jeopardized the mother, fetus or infant, or required intervention to prevent one of the outcomes, or was described as Guillain-Barré Syndrome. Association was determined by a clinician licensed to diagnose and listed on the site's FDA Form 1572.
Time Frame: Day 0 through Day 180 after vaccination
Population: All participants receiving vaccination are included in the safety cohort
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: 8 days after vaccination (Days 0-7).
Population: All participants receiving the vaccination are included in the safety cohort.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants
  Pain | 19 | 23 | 16 | 5 | 9 | 9
  Tenderness | 29 | 37 | 33 | 8 | 11 | 8
  Swelling | 5 | 1 | 0 | 1 | 0 | 1

6. Secondary Outcome: Hemagglutination Inhibition Assay (HAI) Geometric Mean Titer (GMT) Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine at 6 Months After Vaccination
Description: Blood was collected for HAI assay at approximately Day 180 following vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: Day 180 (approximately 6 months after vaccination)
Population: Subjects who received vaccination and contributed blood samples from which valid results were reported are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 45 | 43 | 43 | 15 | 16 | 13
Titer
  B Antigen | 19.7 [14.1 to 27.4] | 23.1 [17.2 to 31.1] | 23.1 [15.6 to 34.4] | 24.1 [11.9 to 48.6] | 18.3 [10.4 to 32.4] | 21.1 [12.8 to 34.7]
  H3N2 Antigen | 47.4 [30.9 to 72.6] | 58.0 [37.5 to 89.5] | 43.4 [27.8 to 67.6] | 40.0 [22.4 to 71.5] | 54.2 [28.4 to 103.4] | 61.3 [22.4 to 167.4]
  H1N1 Antigen | 82.5 [56.9 to 119.6] | 121.6 [88.7 to 166.9] | 85.3 [52.5 to 138.7] | 115.8 [71.8 to 186.8] | 108.3 [57.6 to 203.9] | 208.9 [96.2 to 453.4]

7. Secondary Outcome: Number of Participants With 4-fold or Greater Serum HAI Antibody Titer Increases Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine at 6 Months After Vaccination
Description: Blood was collected from all participants at 180 days after vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 10 (the assay's lowest level of detection) and the Day 180 post vaccination titer was 40 or greater, or the Day 0 titer was greater than or equal to 10 and the Day 180 post vaccination titer was an increase by 4-fold or more.
Time Frame: Day 180 (approximately 6 months after vaccination)
Population: Subjects who received vaccination and contributed blood samples from which valid results were reported are included.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 45 | 43 | 43 | 15 | 16 | 13
participants
  B Antigen | 11 | 11 | 11 | 3 | 2 | 1
  H3N2 Antigen | 13 | 11 | 9 | 3 | 4 | 1
  H1N1 Antigen | 26 | 30 | 23 | 8 | 10 | 9

8. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: 8 days after vaccination (Days 0-7).
Population: All participants receiving the vaccination are included in the safety cohort.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants
  Redness | 7 | 4 | 4 | 2 | 0 | 2
  Swelling | 5 | 2 | 0 | 1 | 1 | 1

9. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: 8 days after vaccination (Days 0-7).
Population: All participants receiving the vaccination are included in the safety cohort.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants
  Feverishness | 1 | 1 | 3 | 1 | 1 | 0
  Malaise | 10 | 10 | 13 | 5 | 4 | 2
  Myalgia | 2 | 6 | 5 | 2 | 5 | 2
  Headache | 11 | 17 | 15 | 4 | 5 | 4
  Nausea | 3 | 3 | 1 | 0 | 2 | 0

10. Primary Outcome: Number of Participants Reporting Fever After Vaccination
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 37.8 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 37.8 degrees Celsius or higher on any of the 8 days.
Time Frame: 8 days after vaccination (Days 0-7).
Population: All participants receiving the vaccination are included in the safety cohort.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 46 | 15 | 16 | 13
participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With HAI Antibody Titer of 40 or Greater Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine at 6 Months After Vaccination
Description: Blood was collected from all participants at 180 days after vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. Participants are counted if the titer at the timepoint is 40 or greater.
Time Frame: Day 180 (approximately 6 months after vaccination)
Population: Subjects who received vaccination and contributed blood samples from which valid results were reported are included.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 45 | 43 | 43 | 15 | 16 | 13
participants
  B Antigen - Day 180 | 16 | 19 | 17 | 6 | 6 | 4
  H3N2 Antigen - Day 180 | 28 | 28 | 24 | 11 | 12 | 8
  H1N1 Antigen - Day 180 | 35 | 40 | 34 | 14 | 13 | 12

12. Secondary Outcome: Maternal HAI GMT Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine at Time of Delivery
Description: Maternal blood was collected for HAI assay at time of delivery. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: At time of delivery
Population: Subjects who contributed blood samples at delivery from which valid results were reported are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 44 | 41 | 43
Titers
  B Antigen | 20.0 [14.3 to 27.9] | 24.1 [17.7 to 32.7] | 21.7 [14.5 to 32.4]
  H3N2 Antigen | 46.8 [30.4 to 72.2] | 61.0 [37.8 to 98.5] | 44.1 [28.5 to 68.1]
  H1N1 Antigen | 86.6 [58.8 to 127.4] | 144.6 [99.4 to 210.2] | 88.1 [53.1 to 146.3]

13. Primary Outcome: Hemagglutination Inhibition Assay (HAI) Geometric Mean Titer (GMT) Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 28 days following vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: Day 0 prior to and Day 28 following vaccination
Population: Subjects who received vaccination and contributed blood samples from which valid results were reported are included. One subject who did not meet eligibility criteria was not included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 45 | 15 | 16 | 13
Titers
  B Antigen - Day 0 | 9.4 [7.5 to 11.8] | 10.6 [8.0 to 14.1] | 8.7 [6.6 to 11.4] | 13.2 [7.0 to 24.8] | 11.4 [7.0 to 18.6] | 23.5 [12.9 to 42.6]
  B Antigen - Day 28 | 36.7 [27.4 to 49.1] | 43.9 [33.3 to 57.8] | 33.8 [23.3 to 48.8] | 40.0 [21.3 to 75.3] | 35.1 [18.6 to 66.3] | 42.2 [27.3 to 65.2]
  H3N2 Antigen - Day 0 | 18.6 [12.6 to 27.4] | 20.6 [12.9 to 32.9] | 17.4 [11.7 to 25.8] | 25.2 [11.9 to 53.3] | 23.8 [10.5 to 53.7] | 42.2 [14.0 to 126.9]
  H3N2 Antigen - Day 28 | 81.2 [53.4 to 123.3] | 105.6 [72.0 to 154.8] | 82.5 [54.7 to 124.5] | 69.6 [34.1 to 142.2] | 134.5 [82.0 to 220.8] | 93.9 [32.6 to 269.9]
  H1N1 Antigen - Day 0 | 16.1 [10.8 to 24.0] | 18.8 [12.4 to 28.4] | 18.5 [12.2 to 28.1] | 31.7 [15.7 to 64.3] | 14.8 [8.6 to 25.3] | 27.5 [12.9 to 58.7]
  H1N1 Antigen - Day 28 | 177.0 [129.0 to 242.8] | 340.3 [260.9 to 443.9] | 183.8 [114.3 to 295.6] | 291.8 [166.8 to 510.5] | 334.2 [187.2 to 596.6] | 417.8 [185.5 to 940.8]

14. Primary Outcome: Number of Participants With 4-fold or Greater Serum HAI Antibody Titer Increases Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine
Description: Blood was collected from all participants prior to vaccination as well as 28 days after vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 10 (the assay's lowest level of detection) and the Day 28 post vaccination titer was 40 or greater, or the Day 0 titer was greater than or equal to 10 and the Day 28 post vaccination titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 28 after vaccination
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 45 | 15 | 16 | 13
participants
  B Antigen | 19 | 23 | 14 | 4 | 5 | 2
  H3N2 Antigen | 24 | 26 | 21 | 5 | 10 | 3
  H1N1 Antigen | 37 | 39 | 32 | 9 | 14 | 10

15. Primary Outcome: Number of Participants With HAI Antibody Titer of 40 or Greater Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine
Description: Blood was collected from all participants prior to vaccination as well as 28 days after vaccination. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. Participants are counted if the titer at the timepoint is 40 or greater.
Time Frame: Day 0 prior to and Day 28 after vaccination
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Number analyzed (Participants) | 48 | 45 | 45 | 15 | 16 | 13
participants
  B Antigen - Day 0 | 5 | 7 | 5 | 4 | 3 | 6
  B Antigen - Day 28 | 26 | 32 | 19 | 10 | 9 | 9
  H3N2 Antigen - Day 0 | 15 | 18 | 11 | 7 | 6 | 7
  H3N2 Antigen - Day 28 | 37 | 37 | 34 | 12 | 16 | 8
  H1N1 Antigen - Day 0 | 14 | 15 | 17 | 9 | 3 | 4
  H1N1 Antigen - Day 28 | 46 | 44 | 40 | 15 | 16 | 12

16. Secondary Outcome: Number of Participants With 4-fold or Greater Maternal Serum HAI Antibody Titer Increases Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine at Time of Delivery
Description: Blood was collected from all participants prior to vaccination as well as at time of delivery. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 10 (the assay's lowest level of detection) and the titer was 40 or greater at delivery, or the Day 0 titer was greater than or equal to 10 and the titer was an increase by 4-fold or more at delivery.
Time Frame: Day 0 prior to vaccination and at time of delivery
Population: Subjects who contributed blood samples at delivery from which valid results were reported are included.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 44 | 41 | 43
participants
  B Antigen | 10 | 7 | 9
  H3N2 Antigen | 13 | 14 | 9
  H1N1 Antigen | 26 | 33 | 23

17. Secondary Outcome: Number of Participants With a Maternal Serum HAI Antibody Titer Greater Than or Equal to 40 Against Each Antigen Included in the 2010-2011 Inactivated TIV at Time of Delivery.
Description: Maternal blood was collected for HAI assay at time of delivery. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. Participants are counted if the titer at the timepoint is 40 or greater.
Time Frame: At time of delivery
Population: Subjects who contributed blood samples at delivery from which valid results were reported are included.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 44 | 41 | 43
participants
  B Antigen | 15 | 15 | 14
  H3N2 Antigen | 29 | 29 | 23
  H1N1 Antigen | 34 | 39 | 34

18. Secondary Outcome: HAI GMT Against Each Antigen in the 2010-2011 Seasonal Influenza Trivalent Influenza Vaccine in Cord Blood Collected at Time of Delivery
Description: Cord blood was collected at delivery for HAI assay at time of delivery. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen.
Time Frame: At time of delivery
Population: Subjects from whom cord blood samples were collected at delivery from which valid results were reported are included.
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 41 | 41 | 41
Titers
  B Antigen | 27.1 [19.2 to 38.3] | 32.1 [23.1 to 44.7] | 28.5 [17.5 to 46.4]
  H3N2 Antigen | 58.0 [35.7 to 94.4] | 71.1 [42.2 to 119.8] | 51.5 [30.5 to 87.3]
  H1N1 Antigen | 124.2 [81.6 to 189.0] | 244.2 [176.6 to 337.6] | 135.1 [79.6 to 229.2]

19. Secondary Outcome: Number of Participants With HAI Antibody Titer Greater Than or Equal to 40 Against Each Antigen Included in the 2010-2011 Inactivated TIV in Cord Blood Collected at Time of Delivery.
Description: Cord blood was collected at delivery for HAI assay at time of delivery. The HAI assay was conducted with the three antigens in the 2010-2011 seasonal inactivated TIV: Influenza B antigen, H1N1 antigen, and H3N2 antigen. Participants are counted if the titer at the timepoint is 40 or greater.
Time Frame: At time of delivery
Population: Subjects from whom cord blood samples were collected at delivery from which valid results were reported are included.
Measure: Number; unit: participants
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants
Number analyzed (Participants) | 41 | 41 | 41
participants
  B Antigen | 19 | 23 | 17
  H3N2 Antigen | 27 | 27 | 24
  H1N1 Antigen | 34 | 39 | 33

ADVERSE EVENTS:
Time Frame: Solicited systemic symptoms and injection site reactions were collected for 8 days (Day 0-7) after vaccination. Unsolicited adverse events were collected for 28 days after vaccination. Serious adverse events were collected for 6 months after vaccination.
Description: For events solicited on the Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | Agriflu (Novartis) in Pregnant Participants | Fluarix (GSK) in Pregnant Participants | Fluzone (Sanofi Pasteur) in Pregnant Participants | Agriflu (Novartis) in Non-pregnant Participants | Fluarix (GSK) in Non-pregnant Participants | Fluzone (Sanofi Pasteur) in Non-pregnant Participants
Serious Adverse Events (participants affected / at risk) | 16/48 | 18/45 | 17/46 | 0/15 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 37/48 | 41/45 | 40/46 | 13/15 | 14/16 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Agriflu (Novartis) in Pregnant Participants (N=48) | Fluarix (GSK) in Pregnant Participants (N=45) | Fluzone (Sanofi Pasteur) in Pregnant Participants (N=46) | Agriflu (Novartis) in Non-pregnant Participants (N=15) | Fluarix (GSK) in Non-pregnant Participants (N=16) | Fluzone (Sanofi Pasteur) in Non-pregnant Participants (N=13)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Congenital cerebral cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Pelvic kidney (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Hypothermia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Body temperature fluctuation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Foetal heart rate abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Aqueductal stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) — Reported for infant delivered by pregnant participant
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Agriflu (Novartis) in Pregnant Participants (N=48) | Fluarix (GSK) in Pregnant Participants (N=45) | Fluzone (Sanofi Pasteur) in Pregnant Participants (N=46) | Agriflu (Novartis) in Non-pregnant Participants (N=15) | Fluarix (GSK) in Non-pregnant Participants (N=16) | Fluzone (Sanofi Pasteur) in Non-pregnant Participants (N=13)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 7 (7) | 7 (7) | 3 (3) | 2 (2) | 0 (0)
Vaccination site discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaccination site paraesthesia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) — Solicited as Feverishness
Malaise (General disorders) | 10 (10) | 10 (10) | 13 (13) | 5 (5) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 5 (5) | 2 (2) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 11 (11) | 17 (17) | 15 (15) | 4 (4) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 19 (19) | 23 (23) | 16 (16) | 5 (5) | 9 (9) | 9 (9)
Tenderness (General disorders) | 29 (29) | 37 (37) | 33 (33) | 8 (8) | 11 (11) | 8 (8) — Solicited as a reaction at the vaccination site
Injection site erythema (General disorders) | 7 (7) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Injection site swelling (functional grading) (General disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Solicited based on impact on daily activities
Injection site swelling (measured reaction) (General disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Solicited as a measured value in millimeters

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less